CLINICAL TRIAL: NCT03568149
Title: Ultrasound Evaluation of the Prevalence of Pelvic Congestion Syndrome in Patients With Endometriosis
Brief Title: Pelvic Congestion Syndrome and Endometriosis
Acronym: VES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Mohamed Mabrouk, Principal investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: VES Study
Record Dates: First submitted 2018-06-11; First posted 2018-06-26 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Pelvic Congestive Syndrome; Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: endometriosis: assessment of pain symptoms at first medical examination; assessment of pelvic vascular insufficiency signs.
  Interventions: Procedure: assessment of pain symptoms at first medical examination; Procedure: assessment of pelvic vascular insufficiency signs
- Group B: no endometriosis: assessment of pain symptoms at first medical examination; assessment of pelvic vascular insufficiency signs.
  Interventions: Procedure: assessment of pain symptoms at first medical examination; Procedure: assessment of pelvic vascular insufficiency signs

INTERVENTIONS:
Procedure: assessment of pain symptoms at first medical examination — First medical examination consists of collection of medical history and standard gynecological examination (bimanual gynecological examination and abdominopelvic ultrasounds). Data regarding age, Body Mass Index, ongoing hormone therapy and pelvic pain symptoms, assessed according to Visual Analogue Scale (VAS) (from 0= no pain to 10= unbearable pain), are collected. The presence of perineal or lower limb varices and the presence and localization of evoked pain at bimanual gynecological examination are also evaluated.
Procedure: assessment of pelvic vascular insufficiency signs — Assessment of pelvic vascular insufficiency in conducted using abdominopelvic ultrasounds, according to the following parameters:
  * Ovarian vein diameter <4mm
  * Slow ovarian blood flow (<3cm/sec)
  * Retrograde blood flow
  * Dilated arcuate veins communicating with pelvic varices The presence of pelvic varices is evaluated qualitatively as normal, moderate and serious
  This evaluation includes the study of uterine and ovarian vessels, using different techniques:
  * Standard 2D study, to measure vessels diameter
  * Vascular doppler study, to evaluate flow direction and blood speed
  * 3D color study, for a three- dimensional reconstruction of vessels and a more accurate qualitative assessment of the congestion degree.

SUMMARY:
The pelvic congestion syndrome (PCS) is a complex and multifactorial condition associated with inflammatory and hormonal etiophatogenesis similar to the endometriosis.

Furthermore, both pathologies share same clinical symptoms as chronic pelvic pain and dyspareunia.

Our hypothesis is that PCS prevalence is higher in patients with endometriosis than in those without clinical or ultrasound signs of endometriosis.

DETAILED DESCRIPTION:
Patients undergoing routine gynecological examinations are included in the study.

Patients are divided into 2 groups:

* Group A: with endometriosis
* Group B: without clinical or ultrasound signs of endometriosis This is an observational, monocentric, prospective, exploratory study. The aim is to assess PCS incidence, associated symptoms and ultrasound characteristics in patients with endometriosis and to compare those findings to those of patients who do not present clinical or ultrasound signs of endometriosis.

The study also evaluates the correlation between:

* Type of pain symptoms (dysmenorrhea, chronic pelvic pain, ovulation pain, dyspareunia, dysuria, dyschezia) and PCS
* Pain severity (assessed according to VAS scale from 0= no pain to 10= unbearable pain) and PCS
* Symptoms and ongoing medical treatments
* History of pelvic surgery and PCS.

Ultrasound parameters of pelvic vascular insufficiency are:

* Ovarian vein diameter <4mm
* Slow ovarian blood flow (<3cm/sec)
* Retrograde blood flow
* Dilated arcuate veins communicating with pelvic varices
* The presence of pelvic varices is evaluated qualitatively as normal, moderate and serious

This evaluation includes the study of uterine and ovarian vessels, using different techniques:

* Standard 2D study: it allows to measure vessels diameter
* Vascular doppler study: it allows to evaluate flow direction and blood speed
* 3D color study: it allows a three- dimensional reconstruction of vessels and a more accurate qualitative assessment of the congestion degree.
* Ultrasound images are evaluated independently by two operators.

ELIGIBILITY:
Inclusion Criteria (Group A):

* Obtaining Informed Consent
* Nulliparity
* Clinical or ultrasounds signs of endometriosis

Inclusion Criteria (Group B):

* Obtaining Informed Consent
* Nulliparity

Exclusion Criteria:

* Menopause
* Actual or previous pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing routine gynecological examinations in our center are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of pelvic congestive syndrome in patients with endometriosis | 1 day, first medical examination
  Comparison of pelvic congestive syndrome symptoms and ultrasounds characteristics, assessed by standard gynecological examination (bimanual gynecological examination and gynecological ultrasounds), between patients with endometriosis (Group A) and without clinical or ultrasound signs of endometriosis.

SECONDARY OUTCOMES:
Correlation between type of pain and pelvic congestive syndrome | 1 day, first medical examination
  Evaluation of the type of pain (dysmenorrhea, chronic pelvic pain, ovulation pain, dyspareunia, dysuria, dyschezia) presented by patients with pelvic congestive syndrome.
Correlation between pain severity and pelvic congestive syndrome | 1 day, first medical examination
  Evaluation of a possible correlation between pain severity and the presence of pelvic congestive syndrome. Pain severity is assessed according to Visual Analogue Scale (VAS scale from 0= no pain to 10= unbearable pain).
Correlation between symptoms and ongoing medical treatments | 1 day, first medical examination
  Evaluation of a possible correlation between symptoms and ongoing medical treatments in patients with pelvic congestive syndrome
Correlation between history of pelvic surgery and pelvic congestive syndrome | 1 day, first medical examination
  Evaluation of a possible correlation between history of pelvic surgery and the presence of pelvic congestive syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecology and Physiopathology of Human Reproductive Unit, University of Bologna, S. Orsola-Malpighi Hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No